CLINICAL TRIAL: NCT06363877
Title: Wound Irrigation and Peritoneal Lavage With Diluted Aqueous Povidone-Iodine Compared to Saline to Decrease Surgical Site Infections
Brief Title: Diluted Aqueous Povidone-Iodine Compared to Saline to Decrease Surgical Site Infections
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5220078
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Surgical Site Infection
Keywords: Intraoperative Wound Irrigation; Intraoperative Peritoneal Lavage; Povidone-Iodine; Normal Saline; Exploratory Laparotomy; Clean Contaminated Wounds; Contaminated Wounds
MeSH Terms: conditions — Surgical Wound Infection | interventions — Povidone-Iodine; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Povidone-Iodine Intraoperative Peritoneal Lavage and Intraoperative Wound Irrigation (Experimental): Patients in this arm will undergo combined intraoperative peritoneal lavage and intraoperative wound irrigation with a diluted aqueous povidone-iodine solution.
  Interventions: Drug: Povidone-Iodine
- Normal Saline Intraoperative Peritoneal Lavage and Intraoperative Wound Irrigation (Active Comparator): Patients in this arm will undergo combined intraoperative peritoneal lavage and intraoperative wound irrigation with a normal saline solution.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Povidone-Iodine — Peritoneal lavage: With the fascia open, the peritoneum will be washed out with 1L of dilute aqueous povidone-iodine solution allowing the solution to sit in the peritoneum for 2 minutes. This is followed by suctioning of the povidone-iodine solution then wash-out with 2L of normal saline followed by suctioning of the normal saline.
  Wound Irrigation: With the fascia closed, the wound will be irrigated with 500mL povidone-iodine solution, suctioned, then washed-out with 500 mL normal saline.
  Arms: Povidone-Iodine Intraoperative Peritoneal Lavage and Intraoperative Wound Irrigation
Drug: Normal Saline — Peritoneal lavage: With the fascia open, the peritoneum will be washed out with 1L of normal saline allowing the solution to sit in the peritoneum for 2 minutes. This is followed by suctioning of the solution, wash-out with 2L of normal saline, followed by suctioning of the normal saline.
  Wound Irrigation: With the fascia closed, the wound will be irrigated with 500mL normal saline solution, suctioned, then washed-out with 500 mL normal saline.
  Arms: Normal Saline Intraoperative Peritoneal Lavage and Intraoperative Wound Irrigation

SUMMARY:
This is a multicenter randomized controlled trial of 1100 patients to evaluate the superiority of combined intraoperative wound irrigation with intraoperative peritoneal lavage with dilute aqueous povidone-iodine compared to normal saline in male and female patients between the ages of 18 and 80 years old undergoing emergency laparotomies with Centers for Disease Control (CDC) class 2 and 3 wounds.

DETAILED DESCRIPTION:
The main objective is stated in the Brief Summary. The secondary objective is to determine the safety and adverse events of povidone-iodine compared to normal saline for irrigation in patients undergoing emergency laparotomies for CDC class 2 and 3 wounds.

The main questions this study aims to answer are:

* Does combined intraoperative wound irrigation with intraoperative peritoneal lavage with dilute aqueous povidone-iodine decrease surgical site infections?
* Is combined intraoperative wound irrigation and intraoperative peritoneal lavage with dilute aqueous povidone-iodine safe to use compared to normal saline?
* Are there any adverse effects of combined intraoperative wound irrigation and intraoperative peritoneal lavage with dilute aqueous povidone-iodine usage on CDC class 2 and 3 wounds compared to normal saline?

Subjects will be followed over 18 months with follow-up of each patient up to 30 days postoperatively. Randomization of patients will occur prior to going to beginning the emergency laparotomy.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years of age
* undergoing an exploratory laparotomy for Centers for Disease Control class II and III wounds

Exclusion Criteria:

* Pregnancy
* Preoperative abdominal wall skin/soft tissue infection
* Iodine allergy
* Patients unlikely to survive beyond 30 days
* Patients with mesh placement or placement of a foreign body except for drains

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection | Between date of initial operation and post-operative follow up visit (up to 30 days post-operatively)
  Subjects in each study arm will be assessed for presence of surgical site infection using a composite measurement based on the CDC/NHSN Guidelines for Surgical Site Infection (SSI) Event (January 2024).
  The presence of one or more of the following will constitute a surgical site infection:
  1. purulent drainage from the superficial incision, deep incision or the drain in an organ/space
  2. organism(s) identified from an aseptically-obtained specimen from the superficial incision, subcutaneous tissue, deep soft tissues, or fluid or tissue in the organ space by a culture or nonculture based microbiologic testing method
  3. an incision that is deliberately opened by a provider AND patient has at least one of the following signs or symptoms: localized pain or tenderness; localized swelling; erythema; or heat
  4. an abscess or other evidence of infection involving the deep incision or organ/space detected on gross anatomical exam, histopathologic exam, or imaging test

SECONDARY OUTCOMES:
Readmission | Between date of surgery and 30 days post-operatively
  Subjects in each study arm will be assessed for the number of times the subject has been readmitted into the hospital for any cause. This will be tracked by chart review and follow-up until 30 days after the initial operation.
Return to the Operating Room | Between date of surgery and 30 days post-operatively
  Subjects in each study arm will be assessed for the number of times the subject returns to the operating room for any cause. This will be tracked throughout the hospital stay and post-discharge by chart review and follow-up until 30 days after the initial operation.
Ileus | Between date of surgery and 30 days post-operatively
  Subjects in each study arm will be assessed for the development of an ileus. This will be diagnosed by lack of bowel function, physical examination (i.e. abdominal distention, tympany) and KUB x-ray to assess for distended loops of bowel with no transition point identified.
Small Bowel Obstruction | Between date of surgery and 30 days post-operatively
  Subjects in each study arm will be assessed for the development of a small bowel obstruction. This will be diagnosed by lack of bowel function, physical examination (i.e. abdominal distention, tympany) and KUB x-ray to assess for distended loops of bowel with a transition point identified. Additional testing including an upper gastrointestinal series (e.g. small bowel follow through) can be used in a case-by-case if medically necessary for diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University Health, Loma Linda, California, United States